CLINICAL TRIAL: NCT04801719
Title: Endoluminal Radiofrequency Ablation of Tumors Affecting the Bile Ducts
Brief Title: Endoluminal Radiofrequency Ablation for the Treatment of Malignant Biliary Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Tomas Andrasina, Tomáš Andrašina, MD, PhD; Assistant professor, Head of Non-vascular interventions and Computed Tomography of the Department of Radiology and Nuclear Medicine, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNBKRNM0002
Record Dates: First submitted 2021-03-09; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Radiofrequency Ablation; Biliary Tract Cancer; Stent Complication; Brachytherapy
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Intervention Model Description: Two study arms with histologically proven malignant biliary stenosis treated either by endoluminal radiofrequency ablation with subsequent metal stent insertion or metal stent insertion only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm - endoluminal RFA (Experimental): standard treatment protocol for malignant biliary stenosis + endoluminal RFA prior metal stent insertion
  Interventions: Device: Habib™ EndoHPB; Boston Scientific, US; former EMcision Ltd., UK
- Control arm (No Intervention): standard treatment protocol for malignant biliary stenosis which includes metal stent insertion

INTERVENTIONS:
Device: Habib™ EndoHPB; Boston Scientific, US; former EMcision Ltd., UK — Randomised patients in selected arm received endoluminal RFA by 8F catheter (Habib™ EndoHPB; Boston Scientific, US; former EMcision Ltd., UK) before stenting procedure. Repeated ablations were processed through stenotic areas of bile ducts (10W, 90-120s, Rita 1500, Angiodynamics Ltd), all drained biliary tracts were used for introducing catheter and performance of ablation. Ablation procedure was followed with uncovered self-expandable metal stent insertion.
  Arms: Experimental arm - endoluminal RFA

SUMMARY:
The rationale of the study is to explore the safety and efficacy of endoluminal radiofrequency ablation prior metal stent insertion in patiens with malignant biliary stenosis.

DETAILED DESCRIPTION:
The aim of this randomized study was to analyze survival rate in patients with malignant biliary obstruction treated with metal stent insertion with or without previous endoluminal radiofrequency ablation (RFA). Secondary endpoint was to analyze metal stent patency rate and survival rate in the subgroup of infiltrative hilar cholangiocarcinomas standardly treated by brachytherapy and metal stenting.

All patients underwent percutaneous cholangiography followed by transhepatic drainage, all patients underwent histopathologic verification of the stenosis.

Randomised patients in selected arm received endoluminal RFA by 8F catheter (Habib™ EndoHPB; EMcision Ltd., London, UK) before stenting procedure. Repeated ablations were processed through stenotic areas (10W, 90-120s, Rita 1500, Angiodynamics Ltd), all drained biliary tracts were used for introducing catheter and performance of ablation.

In experimental group ablation procedure was followed with uncovered self-expandable metal stent insertion.

Brachytherapy procedure (performed in case of cholangiocarcinoma as institutional treatment standard) was performed through 5F applicator by after loading system of iridium radiation source (HDR brachytherapy, applicator temporarily placed into a drain for 3-4 days). Prescribed dose was 15-24Gy at distance of 1.0cm in 3-4 fractions.

Analyzed characteristics:

Specific therapeutic procedures e.g. systemic chemotherapy, brachytherapy indicated by multidisciplinary tumor board were recorded. Laboratory tests were evaluated withing 24 hours before and after the RFA (AMS, INR, APTT, GMT, total bilirubin, ALP, ALT, AST). The time of initial diagnosis, drainage procedures, ablation and stenting were referred to patient survival. Patients underwent repeated ambulatory follow-up in 3months period (dedicated ultrasound performed by interventional radiologist, in case of bilirubin and obstructive enzymes elevation intensified follow up was performed). Patients time of death was gathered from record of central database of insured persons or from hospital information system. Procedural complications were graded in consensus by interventional radiologists and oncologist according to Common Terminology Criteria for Adverse Events.

Primary stent patency:

Stent patency was defined as the duration from the insertion of the stent until the date of closure. If the cause of death was directly related to stent failure, the date of death was defined as time of stent closure. If no stent failure occurred (i.e. the absence of increased total serum bilirubin levels or the absence of dilation of intrahepatic bile ducts on CT or US examination even if total serum bilirubin level was increased), stent patency was considered as censored at the date of death or at the end of the study period.

Statistical methods:

Analyses were performed using IBM SPSS Statistics 23 (IBM Corporation, Armonk, NY, USA). Basic characteristics were summarized by absolute and relative frequencies and compared using Fisher's exact test (categorical variables), continuous characteristics compared using the Mann-Whitney test. Survival parameters were evaluated by Kaplan-Meier methodology, differences in survival were evaluated by log-rank test. Relationships between survival parameters and endoluminal biliary pathway ablation prior to stent insertion were modelled using one-dimensional Cox regression models and described using a risk ratio (HR) of 95% CI for HR and a p-value corresponding to the relevant regression coefficient. The level of statistical significance in all analyses was set at α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* histologically verified malignant stenosis of bile ducts
* indication of implantation of SEMS by multidisciplinary indication committee
* signed informed consent

Exclusion Criteria:

* life expectancy of less than 3 months
* Karnofsky performance status of <80%
* history or concomitant treatment with intraarterial oncologic therapies (eg, hepatic arterial infusion, chemoembolization)
* ongoing infections resistant to antibiotic therapy
* clinical or biochemical signs of liver or renal failure
* INR ≥ 1.3, serum albumin ≤ 35 g/l, haemoglobin ≤ 100 g/l, serum creatinine ≥ 200μmol/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-01-04 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Stent patency | up to month 36 or death of the patient
  Analysis of metal stent patency since insertion in both study arms (measured in months, Kaplan-Meier estimate).
Overall survival | up to month 36 or death of the patient
  Analysis of overall survival since the diagnosis, initial drainage, and metal stent insertion in both study arms (measured in months, Kaplan-Meier estimate).

SECONDARY OUTCOMES:
Complications of endoluminal RFA of biliary tract | up to day 30
  Procedural complications were graded in consensus by interventional radiologists and oncologist according to Common Terminology Criteria for Adverse Events v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Tomáš Andrašina, MD, Principal Investigator — Brno University Hospital
Locations (1):
- Brno University Hospital, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No